CLINICAL TRIAL: NCT01635907
Title: A Phase 2 Study of Dovitinib in Adults With Advanced Malignant Pheochromocytoma or Paraganglioma
Brief Title: Dovitinib in Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 23811
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Advanced Metastatic Paraganglioma; Advanced Metastatic Pheochromocytoma; Recurrent Paraganglioma; Recurrent Pheochromocytoma; Unresectable Paraganglioma; Unresectable Pheochromocytoma
MeSH Terms: conditions — Paraganglioma; Pheochromocytoma | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dovitinib (Experimental)
  Interventions: Drug: Dovitinib

INTERVENTIONS:
Drug: Dovitinib

SUMMARY:
This study is being conducted to evaluate whether the investigational drug Dovitinib, can shrink or slow the growth of cancer in patients with certain types of neuroendocrine tumors. This study will also further evaluate the safety of this drug.

DETAILED DESCRIPTION:
This investigator-initiated study is being conducted to evaluate whether the investigational drug, Dovitinib, can shrink or slow the growth of cancer in patients with certain types of neuroendocrine tumors (advanced malignant pheochromocytoma or paraganglioma). The primary endpoint will be response rate (Complete + Partial Response) determined by RECIST v 1.1. 25 subjects will be enrolled on this study at the University of Pennsylvania.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced, metastatic, recurrent or unresectable paraganglioma or pheochromocytoma. Pathology report or pathology slides (H&E) confirming histological diagnosis must be available at the time of enrollment.
* Must have measurable disease by RECIST v1.1.
* ECOG performance status 0, 1, 2
* Age greater or equal to 18 years old
* Adequate laboratory results; negative pregnancy test (females of childbearing potential)
* Patients who give a written informed consent obtained according to institutional guidelines

Exclusion Criteria:

* Patients with known untreated brain metastases are excluded. Patients having a history of brain metastasis that have been previously irradiated or resected greater than 3 months prior to enrollment and are clinically and radiographically stable will be considered for enrollment.
* Patients with another primary malignancy within 3 years prior to starting study drug, with the exception of adequately treated in-situ carcinoma of the uterine cervix, or skin cancer (such as basal cell carcinoma, squamous cell carcinoma, or non-melanomatous skin cancer)
* Patients who have received the last administration of an anticancer therapy including chemotherapy, immunotherapy, hormonal therapy and monoclonal antibodies (but excluding nitrosurea, mitomycin-C, targeted therapy and radiation) less than or equal to 4 weeks prior to starting study drug, or who have not recovered from the side effects of such therapy
* Patients who have received the last administration of nitrosurea or mitomycin-C less than or equal to 6 weeks prior to starting study drug, or who have not recovered from the side effects of such therapy
* Patients who have received bevacizumab, sunitinib, sorafenib, or pazopanib less than or equal to 2 weeks prior to starting study drug, or who have not recovered (grade 1) from the side effects of these therapies.
* Patients who have had radiotherapy less than or equal to 4 weeks prior to starting study drug, or less than or equal to 2 weeks prior to starting study drug in the case of localized radiotherapy (e.g. for analgesic purpose or for lytic lesions at risk of fracture), or who have not recovered from radiotherapy toxicities
* Patients who have had therapeutic radiolabeled MIBG or other systemic radiolabeled therapy less than or equal to 4 weeks prior to starting study drug,
* Patients who have undergone major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury less than or equal to 4 weeks prior to starting study drug, or patients who have had minor procedures, percutaneous biopsies or placement of vascular access device 1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury
* Patients with any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study (i.e. impaired cardiac function or clinically significant cardiac diseases, etc).
* Pregnant or breastfeeding women or any subjects who refuse to use protocol required contraception
* Patients unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-06; Primary Completion 2016-03 (Actual); Study Completion 2016-04-11 (Actual)

PRIMARY OUTCOMES:
to determine the objective response rate of dovitinib in subjects with advanced malignant pheochromocytoma or paraganglioma | 2 years
  using RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Keefe, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States